CLINICAL TRIAL: NCT00921063
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, 5-Week Trial To Assess The Efficacy And Safety Of PD 0332334 Compared To Placebo And Alprazolam Extended-Release In Patients With Generalized Anxiety Disorder
Brief Title: A 5-Week Trial Of PD 0332334 And Alprazolam Extended Release Compared To Placebo In Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5361007
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — imagabalin; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PD 0332334 250 mg (Experimental)
  Interventions: Drug: PD 0332334
- PD 0332334 100 mg (Experimental)
  Interventions: Drug: PD 0332334
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Alprazolam extended release (Active Comparator)
  Interventions: Drug: Alprazolam extended release

INTERVENTIONS:
Drug: PD 0332334 — 250 mg capsule, BID for 4 weeks
  Other Names: imagabalin
  Arms: PD 0332334 250 mg
Drug: PD 0332334 — 100 mg capsule, BID for 4 weeks
  Arms: PD 0332334 100 mg
Drug: placebo — 0 mg capsule, BID for 4 weeks
  Arms: placebo
Drug: Alprazolam extended release — 1 mg capsule, BID for 4 weeks
  Other Names: Xanax XR
  Arms: Alprazolam extended release

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of PD 0332334 compared to placebo in the treatment of Generalized Anxiety Disorder in an adult population

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females with a diagnosis of Generalized Anxiety Disorder (GAD) (Diagnostic and Statistical Manual-IV [DSM-IV], 300.02).
* HAM-A Total Score ≥20 and item #1 on the HAM-D (depressed mood score) ≤2 at both Screening and Baseline/Randomization.

Exclusion Criteria:

* Current diagnoses (within the 6 months) of Major Depressive Disorder; Obsessive Compulsive Disorder; Panic Disorder; Posttraumatic Stress Disorder; Anorexia; Bulimia; Caffeine-induced anxiety disorder;
* Any of the following past or current diagnoses: Schizophrenia; Psychotic Disorder; Delirium, Dementia, Bipolar or Schizoaffective Disorder; Cyclothymic Disorder; Dissociative Disorders; Antisocial or borderline personality disorder
* Current use of psychotropic medications (i.e., drugs normally prescribed for depression, mania, anxiety, insomnia, or psychosis) that could not be discontinued 2 weeks prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2005-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
HAM-A Total Score | 4 weeks

SECONDARY OUTCOMES:
HAM-A total score at week 1, 2 and 4 | 1. 2. ands 4 weeks
HAM-A somatic and psychic subscales | 1, 2, and 4 weeks
HAM-A responders | 4 weeks
HAM-A sustained responders | Week 1 through week 4
DAS-A (daily assessment of symptoms of anxiety) and GA-VAS (VAS scale for global anxiety) | Day 2 through day 7
CGI-I (Clinical Global Impression of Improvement) and PGI-I (Patient Global Impression of Change) | 1 and 4 weeks
HAM-D total score | 1 and 4 weeks
Sheehan Disability Score (SDS) | 4 weeks
Treatment Satisfaction Questionaire for Medication | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361007&StudyName=A%205-Week%20Trial%20Of%20PD%200332334%20And%20Alprazolam%20Extended%20Release%20Compared%20To%20Placebo%20In%20Patients%20With%20Generalized%20Anxiety%20Disorder